CLINICAL TRIAL: NCT05505955
Title: A Phase I Study to Evaluate Safety, Tolerability, Pharmacokinetics/Pharmacodynamics of Single and Multiple Dose of HRS-5965 Tablets in Healthy Subjects, and the Food Effect on Pharmacokinetics, and Pharmacokinetics in Subjects With Impaired Renal Function
Brief Title: Study of HRS-5965 in Healthy Subjects and Subjects With Renal Insufficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chengdu Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-5965-101
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Glomerulonephritis
MeSH Terms: conditions — Glomerulonephritis

STUDY DESIGN:
Intervention Model Description: Single-dose and multi-dose, dose escalation, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1 (Experimental): single ascending dose, randomized, double-blind study，with 6 dose groups preset, of which 1 group will be administered under fasted and fed conditions. The food impact study consisted of 10 subjects, 8 of whom received HRS-5965 tablets and 2 of whom received placebo. The remaining cohorts required 8 subjects each, with 6 receiving HRS-5965 tablets and 2 receiving placebo.
  Interventions: Drug: HRS-5965; Drug: Placebo
- Part 2 (Experimental): Multiple ascending dose, randomized, double-blind study，with 4 dose groups preset; Each dose group consisted of 8 healthy adult subjects randomly assigned 6:2 to HRS-5965 tablets or placebo.
  Interventions: Drug: HRS-5965; Drug: Placebo
- Part 3 (Experimental): an open-label, nonrandomized, single-dose study to evaluate the effect of severe renal impairment (RI) on the safety, tolerability, pharmacokinetics, and pharmacodynamics of HRS -5965 compared to demographically-matched healthy participants with normal renal function. Subjects took HRS5965 tablets.
  Interventions: Drug: HRS-5965

INTERVENTIONS:
Drug: HRS-5965 — Subjects took HRS5965 tablets in Part 1, Part 2 and Part 3.
Drug: Placebo — Subjects took Placebo in Part 1 and Part 2.
  Arms: Part 1; Part 2

SUMMARY:
The trial is the first human trial. The safety, tolerability, PK and PD of HRS-5965 tablets will be evaluated in healthy subjects and subjects with impaired renal function. The study was divided into three parts:

Part 1: single ascending dose, randomized, double-blind study，with 6 dose groups preset, of which 1 group will be administered under fasted and fed conditions; Part 2: Multiple ascending dose, randomized, double-blind study，with 4 dose groups preset; Part 3: an open-label, nonrandomized, single-dose study to evaluate the effect of severe renal impairment (RI) on the safety, tolerability, pharmacokinetics, and pharmacodynamics of HRS -5965 compared to demographically-matched healthy participants with normal renal function.

ELIGIBILITY:
Inclusion Criteria:

- Healthy subjects study

1. Healthy male or female, age ≥ 18 years old and ≤ 70 years old (on the day of signing the informed consent);
2. 18.5kg/m2 ≤BMI<30 kg/m2, and the weight of men should be ≥ 50kg, and that of women should be ≥ 45kg.

Study on subjects with renal insufficiency

1. Age ≥ 18 years old and ≤ 70 years old (on the day of signing the informed consent), both men and women can;
2. 18.5kg/m2≤BMI<30 kg/m2；
3. The estimated glomerular filtration rate of subjects with chronic renal insufficiency conforms to 15 ≤ EGFR < 30 ml/min/1.73m2 (calculated according to CKD-EPI formula, see Appendix 2 of the scheme).

Exclusion Criteria:

- Healthy subjects study

1. The researcher has determined that there may be diseases or medical conditions that affect the absorption, distribution, metabolism and excretion of drugs or reduce compliance;
2. The estimated glomerular filtration rate conforms to EGFR < 90 ml/min/1.73m2 (calculated according to CKD-EPI formula, see Appendix 2 of the scheme);
3. According to the judgment of the researcher, any physiological or psychological disease or condition that may increase the risk of the test, affect the subject's compliance with the protocol, or affect the subject's completion of the test.

Study on subjects with renal insufficiency

1. Those who received renal replacement therapy within 12 weeks before screening; Or the two tests in the screening period indicate that the renal function is unstable (the results in the screening period meet the diagnostic criteria of 2012 KDIGO acute renal injury, or the changes that do not meet the above criteria but are judged to be clinically significant by the researcher. If there are reasonable reasons, the third test is allowed, and the interval between two consecutive tests should be more than 3 days but not more than 7 days);
2. According to the judgment of the researcher, the subject has any of the following: in the state of progression or prognosis of disease (including primary renal disease, complications and other complications); The treatment plan needs to be adjusted at any time; Any physical or mental disease or condition that may increase the risk of the test, affect the subject's compliance with the protocol, or affect the subject's completion of the test.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2022-10-08 (Actual); Primary Completion 2023-11-03 (Actual); Study Completion 2023-11-03 (Actual)

PRIMARY OUTCOMES:
The incidence and severity of adverse events to assess safety and tolerability | up to 24 days

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) on Day 1 for Part 1 and Part 3 | Pre-dose to 144 hours post-dose
Peak plasma concentration (Cmax) on Day 1 for Part 1 and Part 3 | Pre-dose to 144 hours post-dose
Time to maximum plasma concentration (Tmax) on Day 1 for Part 1 and Part 3 | Pre-dose to 144 hours post-dose
• Area under the plasma concentration versus time curve (AUC) on Day 1 and Day 10 for Part 2 | Pre-dose to 144 hours post-dose
Peak plasma concentration (Cmax) on Day 1 and Day 10 for Part 2 | Pre-dose to 144 hours post-dose
Time to maximum plasma concentration (Tmax) on Day 1 and Day 10 for Part 2 | Pre-dose to 144 hours post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated hospital of QingDao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xu Y, Tian F, Ren H, Yu X, Chen X, Ye K, Sun F, Fang L, Li Y, Ban R, Jiang X, Wang C, Ma Y, Kuang F, Li X, Zhang Z, Ye C, Hu M, He F, Shu C, Zou Y, Huang R, Shen K, Xing G, Cao Y. HRS-5965, a small-molecule factor B inhibitor, in healthy participants and participants with renal insufficiency: A first-in-human, phase 1 trial. Med. 2025 Aug 8;6(8):100698. doi: 10.1016/j.medj.2025.100698. Epub 2025 May 15. PMID 40378845